CLINICAL TRIAL: NCT03069170
Title: Safety and Efficacy of Immuno-modulation and Autologous Bone Marrow-Derived Stem Cell Transplantation for the Treatment of Multiple Sclerosis.
Brief Title: Autologous Bone Marrow Derived Stem Cells for the Treatment of Multiple Sclerosis.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stem Cells Arabia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA-MS1
Record Dates: First submitted 2017-02-25; First posted 2017-03-03 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2019-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stem Cells (Experimental): Intravenous administration of purified autologous bone marrow-derived stem cells.
  Interventions: Biological: Stem Cell Transplantation
- Stem Cell Transplantation (Experimental): Intrathecal administration of purified autolgous bone-marrow derived stem cells.
  Interventions: Biological: Stem Cell Transplantation

INTERVENTIONS:
Biological: Stem Cell Transplantation — Intravenous and Intrathecal injections of purified autologus bone marrow-derived stem cells.

SUMMARY:
Until now, there is no effective approach to stop the progression of multiple sclerosis and stimulate re-myelination. Autologous stem cell transplantation shows hope and is quickly developing as an alternative therapy. We propose the use of autologous bone marrow-derived specific stem cell populations and mesenchymal stem cell transplantation (BM-MSC) associated with immuno-modulation to treat patients with relapsing-remitting MS (RRMS).

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune de-myelinating disease in which the myelin sheaths of nerve cells in the central nervous system are damaged.This damage disrupts the ability of parts of the nervous system to communicate, resulting in a range of signs and symptoms, including physical, mental, and psychiatric issues. To date, There is no known cure for multiple sclerosis. Treatments attempt to improve function after an attack and prevent new attacks.

Stem cells possess strong immunomodulatory properties that are shown to play a role in the maintenance of peripheral tolerance and in the control of autoimmunity and that may stimulate repair and regeneration of lesion. Clinical studies have shown that stem cells can be safely harvested and do not form tumors. Most of human stem cell trials have focused on clinical applications for haematopoietic stem cells (HSC), mesenchymal stem cells (MSC), or both. When administered intravenously they have an immune inhibitory effect that can ameliorate animal autoimmune diseases. MSC transplantation significantly improves clinical outcome in experimental allergic encephalitis (EAE). When administered intravenously, MSC may migrate to inflammatory brain lesions and promote survival of nervous cells. Hence, MSC have become the focus of studies as a potential cell therapy for stimulating neuro-protection in human neurodegenerative diseases such as MS.

We propose a safety and efficacy trial of a intravenous and intrathecal injections of autologous bone marrow-derived stem cells into patients with MS.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting MS (RRMS) patients
* Age 18-50 years
* Disease duration >= 2 and <= 10 years
* EDSS: 3.0 - 6.5

Exclusion Criteria:

* RRMS not fulfilling inclusion criteria
* SPMS or PPMSTreatment with any immunosuppressive therapy
* Treatment with interferon-beta or glatiramer acetate within the 30 days prior to transplantation
* Treatment with corticosteroids within the 30 days prior to transplantation
* Relapse occurred during the 60 days prior to transplantation
* History of cancer or clinical or laboratory results indicative of severe systemic diseases, including infection for HIV, Hepatitis B or C
* Pregnancy or risk of pregnancy/ lactation
* Current treatment with an investigational therapy
* Inability to give written informed consent in accordance with research ethics board guidelines

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2020-09 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness assessment by MRI | 6 months
Safety assessment by physical examination, vital signs, analytical results, electrocardiograph monitoring, and Expanded Disability Status Scale (EDSS) | 12 months

SECONDARY OUTCOMES:
Change in Quality of life by Multiple Sclerosis Quality of Life (MSQOL-54) | 6 months
Axonal effect by Optical coherence tomography (OCT) | 6 months
Immunology: Dosing of G, A and M immunoglobulins, and complement factors C3 and C4 | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Stem Cells Arabia, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided